CLINICAL TRIAL: NCT01516164
Title: A Comparison of the Ease of Tracheal Intubation Using a McGrath MAC Laryngoscope and a Standard MacIntosh Laryngoscope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Tayside (Other Government)
Responsible Party: Principal Investigator, Dr Claire Wallace, Dr Claire Wallace SpR Anaesthetics, NHS Tayside
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011AN04
Record Dates: First submitted 2012-01-19; First posted 2012-01-24 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-10

CONDITIONS: Tracheal Intubation
Keywords: Laryngoscopy; Videolaryngoscopy; Ease of Intubation
MeSH Terms: interventions — Laryngoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- MacIntosh (Active Comparator)
  Interventions: Device: Laryngoscopy
- McGrath MAC direct (Active Comparator)
  Interventions: Device: Laryngoscopy
- McGrath MAC indirect (Active Comparator)
  Interventions: Device: Laryngoscopy

INTERVENTIONS:
Device: Laryngoscopy — After establishing full monitoring, inducing general anaesthesia and ensuring paralysis laryngoscopy is performed and the patient's trachea intubated.

SUMMARY:
Videolaryngoscopes offer the potential to make tracheal intubation easier for the anaesthetist and less traumatic for the patient. This study aims to compare the intubation difficulty scores (a validated scoring system for ease of intubation) using the McGrath MAC as a videolaryngoscope, the McGrath MAC only as a direct laryngoscope (without video screen) and the MacIntosh laryngoscopes.

ELIGIBILITY:
Inclusion Criteria:

* Elective procedure requiring oral tracheal tube intubation
* Over 16 years of age
* Airway assessment suggests to the anaesthetist that a standard MacIntosh laryngoscope approach to intubation would be appropriate.

Exclusion Criteria:

* Emergency procedure
* Less than 16 years of age
* Unable to consent
* Requiring Rapid Sequence Induction (a specialised anaesthetic induction technique)
* Predicted difficult intubation
* Not suitable for the standardised induction technique

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2012-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Intubation Difficulty Score | 5 minutes
  The Intubation Difficulty Scale (IDS) is a numerical score based on seven parameters. The scoring of each parameter represents a divergence from an 'ideal' condition and the total score represents a sum divergence from a zero difficulty ideal intubation. The seven parameters are number of supplementary attempts, number of supplementary operators, number and type of alternative techniques used, laryngoscopic grade, subjective lifting force, the use of external laryngeal manipulation and mobility or position of the vocal cords.

SECONDARY OUTCOMES:
Time to intubation | 5 minutes
Number and types of alternative techniques used | 5 minutes
Perception of force used | 5 minutes
Complications | 5 minutes
Ease of intubation | 5 minutes
Failure to intubate | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Claire D Wallace, MBChB, Principal Investigator — NHS Tayside
Locations (1):
- NHS Tayside, Tayside, Tayside, United Kingdom